CLINICAL TRIAL: NCT03011879
Title: China STEMI Care Project Phase 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Chinese Medical Doctor Association (Other)
Responsible Party: Principal Investigator, Yong Huo, Director, Department of Cardiology, Peking University First Hospital
Other Study IDs: CSCAP-2
Record Dates: First submitted 2016-08-27; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: ST-Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Critical Pathways

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — patients under thrombolysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1.STEMI patients with symptom onset within 30 days: First round enrollment of STEMI patients with symptom onset within 30 days
  Interventions: Other: clinical pathway
- 2.STEMI patients with symptom onset within 30 days: Second round enrollment of STEMI patients with symptom onset within 30 days
  Interventions: Other: clinical pathway
- 3.STEMI patients with symptom onset within 30 days: Third round enrollment of STEMI patients with symptom onset within 30 days
  Interventions: Other: clinical pathway

INTERVENTIONS:
Other: clinical pathway

SUMMARY:
The program is to improve STEMI medical care quality in China. With the documents issued by National Health and Family Planning Commission of the People's Republic of China, the program was initialed in at least 200 primary PCI capable hospitals together with hundreds of adjacent non-primary PCI capable hospitals in 15 provinces. STEMI patients with symptom onset within 30 days will be enrolled in 3 periods. In each period with 6-month interval, 30 patients will be enrolled consecutively from each PCI-capable center initially and from non-primary PCI capable hospitals later, thus at least 18,000 STEMI patients from primary PCI capable hospitals will be enrolled and all of them will be followed up for 1 year. Key performance indicators (KPIs) in STEMI care will be collected using both national PCI online registry and a program STEMI online registry database for the purpose of improvement of medical care. Hospital KPIs rank report and problem-based resolution will be feedback to each hospital after data analysis in each period. Comparison of every two cross-sectional data (self) and within one cross-sectional (inter-hospital) data will be used to evaluate the improvement of medical quality.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients with symptom onset within 30 days

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI patients with symptom onset within 30 days
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Referfusion ratio in patients with symptom onset within 12 hours | 12 hours
  Referfusion including primary PCI and thrombolysis is the key strategy in STEMI care
Door-to-ballnoon time in patients with symptom onset within 12 hours | 12 hours
  Door-to-ballnoon time is the key index to evaluate treatment of primary PCI
Door-to-needle time in patients with symptom onset within 12 hours | 12 hours
  Door-to-needle time is the key index to evaluate treatment of thrombolysis
Hospital admission via ambulance ratio | 2 years
Symptom onset to arrive in hospital | 2 years
Bypass ED ratio in patients with symptom onset within 12 hours | 12 hours
Usage of both DAPT, statin, β blocker and ACEI/ARB in patients without contraindication | 3 yeras
  DAPT means dual antiplatelet therapy
In-hospital morbidity | 2 yeras
1-year on time follow-up ratio | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No